CLINICAL TRIAL: NCT03185819
Title: A Double-blind, Randomized, Psychoactive Placebo-controlled, Study to Evaluate the Efficacy and Safety of 3 Fixed Doses (28 mg, 56 mg and 84 mg) of Intranasal Esketamine in Addition to Comprehensive Standard of Care for the Rapid Reduction of the Symptoms of Major Depressive Disorder, Including Suicidal Ideation, in Pediatric Subjects Assessed to be at Imminent Risk for Suicide
Brief Title: Study to Evaluate the Efficacy and Safety of 3 Fixed Doses of Intranasal Esketamine in Addition to Comprehensive Standard of Care for the Rapid Reduction of the Symptoms of Major Depressive Disorder, Including Suicidal Ideation, in Pediatric Participants Assessed to be at Imminent Risk for Suicide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108323; 2016-004422-42 (EudraCT Number); ESKETINSUI2002 (Other: Janssen Research & Development, LLC)
Expanded Access: NCT03829579 (Approved for marketing)
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Midazolam; Esketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Oral Midazolam + Intranasal Placebo (Placebo Comparator): Participants will receive midazolam solution 0.125 milligram per kilogram (mg/kg) orally 2 times per week for 4 weeks and 3 intranasal doses of matched placebo to esketamine.
  Interventions: Drug: Intranasal Placebo; Drug: Midazolam
- Oral Placebo + Esketamine 84 mg (Experimental): Participants will receive intranasal esketamine 84 mg as 3 intranasal doses of esketamine in each nostril (each dose contains 14 mg of esketamine) along with oral placebo 2 times per week for 4 weeks.
  Interventions: Drug: Midazolam Placebo Solution; Drug: Esketamine
- Oral Placebo + Esketamine 56 mg (Experimental): Participants will receive intranasal esketamine 56 mg as 2 intranasal doses of esketamine in each nostril (each dose contains 14 mg of esketamine) along with oral placebo 2 times per week for 4 weeks.
  Interventions: Drug: Midazolam Placebo Solution; Drug: Esketamine
- Oral Placebo + Esketamine 28 mg (Experimental): Participants will receive intranasal esketamine 28 mg as 1 intranasal doses of esketamine in each nostril (each dose contains 14 mg of esketamine) along with oral placebo 2 times per week for 4 weeks.
  Interventions: Drug: Midazolam Placebo Solution; Drug: Esketamine

INTERVENTIONS:
Drug: Intranasal Placebo — Participants will receive placebo as intranasal dose to match intranasal esketamine.
  Arms: Oral Midazolam + Intranasal Placebo
Drug: Midazolam Placebo Solution — Participants will receive placebo as oral dose to match midazolam drug.
  Arms: Oral Placebo + Esketamine 28 mg; Oral Placebo + Esketamine 56 mg; Oral Placebo + Esketamine 84 mg
Drug: Midazolam — Participants will receive midazolam solution 0.125 mg/kg as oral dose to match placebo.
  Arms: Oral Midazolam + Intranasal Placebo
Drug: Esketamine — Participants will receive esketamine at a dose of 28 mg as intranasal solution.
  Arms: Oral Placebo + Esketamine 28 mg
Drug: Esketamine — Participants will receive esketamine at a dose of 56 mg as intranasal solution.
  Arms: Oral Placebo + Esketamine 56 mg
Drug: Esketamine — Participants will receive esketamine at a dose of 84 mg as intranasal solution.
  Arms: Oral Placebo + Esketamine 84 mg

SUMMARY:
The purpose of this study is to assess the efficacy of a single (first) dose of 3 fixed doses of intranasal esketamine {28 milligram (mg), 56 mg, and 84 mg} compared with psychoactive placebo (oral midazolam) in rapidly reducing the symptoms of major depressive disorder (MDD) including suicidal ideation in participants 12 to less than 18 years of age who are assessed to be at imminent risk for suicide.

DETAILED DESCRIPTION:
This study will enroll participants with major depressive disorder (MDD) presenting with suicidal ideation who are assessed to be at imminent risk for suicide. The study will be conducted in 4 phases: a screening evaluation performed within 48 hours prior to Day 1 intranasal dose; a 25-day double-blind treatment phase (Days 1-25); an 8-week initial post-treatment phase (Days 25-81); and a subsequent phase to complete a full 6-month post-treatment follow-up (Days 81-200). Efficacy, safety, pharmacokinetic, biomarker, and pharmacogenomic evaluations will be performed in the study at defined schedule. The duration of the participant's participation will be approximately 29 weeks. If you or a loved one are having thoughts of suicide, please seek immediate medical help. Go to the emergency room or call the National Suicide Prevention Lifeline at 1-800-273-8255.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet diagnostic and statistical manual of mental disorders (5th edition) {DSM-5} diagnostic criteria for major depressive disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the mini international neuropsychiatric interview for children and adolescents (MINI KID)
* Participant must have a children's depression rating scale-revised (CDRS-R) total score of equal or more than (>=) 58 predose on Day 1
* As part of standard of care treatment, participant must agree to be hospitalized voluntarily for a recommended period of 5 days after randomization (may be shorter or longer if clinically warranted in the investigator's opinion)
* As part of the newly initiated or optimized standard of care treatment, participant must agree to take one of the prescribed non-investigational antidepressant medications (fluoxetine, escitalopram, sertraline; and 9-11 years old participants at US-sites only: fluoxetin [preferred], sertraline) at least during the double-blind treatment phase (Day 25)
* As part of standard of care treatment, participant must agree to participate in a specific psychological intervention (individual cognitive behavioral therapy [CBT], interpersonal therapy, family therapy or psychodynamic psychotherapy) at least through the initial 8-week post-treatment follow-up period (Day 81)

Exclusion Criteria:

* Participants has a current DSM-5 diagnosis of bipolar (or related disorders), intellectual disability, autism spectrum disorder, conduct disorder, anorexia nervosa, oppositional defiant disorder, or obsessive compulsive disorder
* Participants currently meets DSM-5 criteria for borderline personality disorder. Participants not meeting full DSM-5 criteria for borderline personality disorder but exhibiting recurrent suicidal gestures, threats, or self-mutilating behaviors should also be excluded
* Participant has a current or prior DSM-5 diagnosis of a psychotic disorder or MDD with psychosis
* Participant meets the DSM-5 severity criteria for moderate or severe substance or alcohol use disorder (except for nicotine or caffeine) within the 6 months before screening. A history (lifetime) of ketamine, phencyclidine (PCP), lysergic acid diethylamide (LSD), or 3, 4-methylenedioxy-methamphetamine (MDMA) hallucinogen-related use disorder is exclusionary
* Participant has a history of seizure disorder

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (51):
- United States (18):
  - Institute of Living/ Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Atlanta Behavioral Research, LLC, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Neuroscience Research Institute, Winfield, Illinois
  - Beacon Medical Group Clinical Research, South Bend, Indiana
  - University of Iowa, Carver College of Medicine, Iowa City, Iowa
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Sheppard Pratt Health System, Baltimore, Maryland
  - CBH Health, Gaithersburg, Maryland
  - State University of New York at Buffalo, Buffalo, New York
  - University North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Hospital, Cincinnati, Ohio
  - University Hospital of Cleveland, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
- Hopital Erasme, Brussels, Belgium
- Brazil (4):
  - Trial Tech Tecnologia em Pesquisas com Medicamentos, Curitiba
  - Hospital Universitario Professor Edgar Santos, Salvador
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo
  - Hospital São Sebastião, Turvo
- Bulgaria (2):
  - Mental Health Center - Rousse, Rousse
  - Multiprofile Hospital for Active Treatment - MHAT Sveta Marina EAD, Varna
- France (6):
  - Hospices Civils de Lyon HCL, Bron
  - CHRU Lille - Hôpital Fontan 1, Lille
  - CHU Nantes, Nantes
  - Hôpital Universitaire Pitié-Salpêtrière, Paris
  - Hopital Sainte Anne, Paris
  - Hôpital Robert Debré, Paris
- Hungary (2):
  - Vadaskert Gyermek es Ifjusagpszichiatriai Korhaz es Szakambulancia, Budapest
  - Szegedi Tudomanyegyetem, Szeged
- Italy (7):
  - Azienda Ospedaliera G. Brotzu, Cagliari
  - OSP RIUNITI-DIP Donna- Bambino, Foggia
  - Ospedale di Merano, Merano
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - IRCCS C. Mondino, Istituto Neurologico Nazionale, Fondazione, Pavia
  - Irccs Burlo-Garofalo, Trieste
- Poland (3):
  - Klinika Psychiatrii Dzieci i Mlodziezy, CM UJ, Krakow
  - Dzieciecy Szpital Kliniczny im Jozefa Polikarpa Brudzinskiego, Warsaw
  - Instytut Psychiatrii i Neurologii Klinika Psychiatrii Dzieci i Mlodziezy, Warsaw
- Spain (8):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Sant Joan de Deu, Esplugues de Llobregat
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Infantil Univ. Nino Jesus, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Hosp. Univ. Central de Asturias, Oviedo
  - Clinica Univ. de Navarra, Pamplona
  - Corporacio Sanitari Parc Tauli, Sabadell

REFERENCES:
- [Derived] Kosik-Gonzalez C, Fu DJ, Chen LN, Lane R, Bloch MH, DelBello M, Moreno C, Drevets WC, Canuso CM. Effect of Esketamine on Depressive Symptoms in Adolescents With Major Depressive Disorder at Imminent Suicide Risk: A Randomized Psychoactive-Controlled Study. J Am Acad Child Adolesc Psychiatry. 2026 Jan;65(1):42-55. doi: 10.1016/j.jaac.2025.02.015. Epub 2025 Mar 7. PMID 40058488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 147 participants were randomized and treated. One participant (randomized to arm "Esketamine 84 mg+Placebo+standard of care [SOC]") was excluded from the efficacy analysis set, safety analysis set, and follow-up analysis set due to Good Clinical Practice (GCP) issue at the site.
Pre-assignment Details: Adolescent participants with major depressive disorder (MDD) who were assessed to be at imminent risk for suicide were enrolled in this study.
Groups:
- Placebo + Midazolam + SOC: In the double blind (DB) phase, participants received 3 intranasal doses of placebo (matched to esketamine nasal spray) using 3 devces, each device at time points 0, 5 and 10 minutes (min) respectively. For each device, 1 spray was administered into each nostril (that is total of 2 sprays/device). An oral solution of midazolam 0.125 milligrams per kilogram (mg/kg) was administered immediately before the first intranasal dose. Study drugs were taken 2 times per week for 4 weeks (on Days 1, 4, 8, 11, 15, 18, 22, and 25). During the study, all participants were treated with Standard of care (SOC): antidepressant treatment (either fluoxetine or escitalopram or sertaline) based on clinical judgement, initiated, or optimized on Day 1 or up to 7 days after first dose of study drug administration (on Day 1), if starting two medications simultaneously was not consistent with local clinical practice, and psychotherapy. After DB treatment phase, participants entered post-treatment follow-up (FU) phase and received no study drug.
- Esketamine 28 mg + Placebo + SOC: In DB phase, participants received 1 intranasal dose of esketamine 28 mg nasal spray using a device, at 0 min, followed by 2 intranasal doses of placebo (matched to esketamine) using 2 devices, 1 at 5 min and another at 10 min, respectively. For each device, 1 spray (esketamine 14 mg/placebo) was administered into each nostril (that is total of 2 sprays = esketamine 28 mg/placebo). Placebo oral solution (matched to midazolam 0.125 mg/kg) was administered immediately before first intranasal dose. Study drugs were taken 2 times per week for 4 weeks (on Days 1, 4, 8, 11, 15, 18, 22, and 25). During study, all participants received SOC: antidepressant treatment (fluoxetine or escitalopram or sertaline) based on clinical judgement, initiated or optimized on Day 1 or up to 7 days after first dose (on Day 1), if starting two medications simultaneously was not consistent with local clinical practice, and psychotherapy. After DB phase, participants entered post-treatment FU phase and received no study drug.
- Esketamine 56 mg + Placebo + SOC: In DB phase, participants received 2 intranasal doses of esketamine 56 mg nasal spray using 2 devices, 1 at 0 min and another at 5 min, followed by 1 intranasal dose of placebo (matched to esketamine) using 1 device at 10 min. For each device, 1 spray (esketamine 14 mg/placebo) was administered into each nostril (that is total of 2 sprays = esketamine 28 mg/placebo). Placebo oral solution (matched to midazolam 0.125 mg/kg) was administered immediately before first intranasal dose. Study drugs were taken 2 times per week for 4 weeks (on Days 1, 4, 8, 11, 15, 18, 22, and 25). During study, all participants received SOC: antidepressant treatment (fluoxetine or escitalopram or sertaline) based on clinical judgement, initiated or optimized on Day 1 or up to 7 days after first dose (on Day 1), if starting two medications simultaneously was not consistent with local clinical practice, and psychotherapy. After DB phase, participants entered post-treatment FU phase and received no study drug.
- Esketamine 84 mg + Placebo + SOC: In DB phase, participants received 3 intranasal doses of esketamine 84 mg nasal spray using 3 devices, each device at 0, 5 and 10 min, respectively. For each device, 1 spray (esketamine 14 mg/placebo) was administered into each nostril (that is total of 2 sprays = esketamine 28 mg/placebo). Placebo oral solution (matched to midazolam 0.125 mg/kg) was administered immediately before first intranasal dose. Study drugs were taken 2 times per week for 4 weeks (on Days 1, 4, 8, 11, 15, 18, 22, and 25). During study, all participants received SOC: antidepressant treatment (fluoxetine or escitalopram or sertaline) based on clinical judgement, initiated or optimized on Day 1 or up to 7 days after first dose (on Day 1), if starting two medications simultaneously was not consistent with local clinical practice, and psychotherapy. After DB phase, participants entered post-treatment FU phase and received no study drug.
Period: Double-Blind Phase: Day 1 to Day 25
Arm/Group | Placebo + Midazolam + SOC | Esketamine 28 mg + Placebo + SOC | Esketamine 56 mg + Placebo + SOC | Esketamine 84 mg + Placebo + SOC
Started | 63 | 29 | 31 | 24
Safety Analysis Set (Safety analysis set included all randomized participants who received at least 1 dose of study medication in the double-blind phase.) | 63 | 29 | 31 | 23
Full Efficacy Analysis Set (The full efficacy analysis set included all randomized participants who received at least 1 dose of double-blind study intervention during the double-blind treatment phase and had both baseline and post-baseline evaluation for the CDRS-R total score.) | 63 | 28 | 31 | 23
Follow-up Analysis Set (The follow-up analysis set included all participants who completed the double-blind phase and either entered the follow-up phase or have provided adverse event data after the double-blind phase.) | 59 | 29 | 29 | 21
Completed | 59 | 29 | 29 | 22
Not Completed | 4 | 0 | 2 | 2
Not completed — Withdrawal by parent/guardian | 0 | 0 | 0 | 1
Not completed — Other | 1 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 1 | 0
Not completed — Subject refused further study treatment | 0 | 0 | 0 | 1
Period: Post-treatment Follow-up: Days 26 to 200
Arm/Group | Placebo + Midazolam + SOC | Esketamine 28 mg + Placebo + SOC | Esketamine 56 mg + Placebo + SOC | Esketamine 84 mg + Placebo + SOC
Started | 59 | 29 | 29 | 21
Completed | 48 | 24 | 21 | 18
Not Completed | 11 | 5 | 8 | 3
Not completed — Withdrawal by parent/guardian | 1 | 0 | 1 | 0
Not completed — Other | 1 | 0 | 3 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Requires treatment with electroconvulsive therapy, transcranial magnetic stimulation, ketamine | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 2 | 0
Not completed — Physician Decision | 2 | 0 | 2 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 2
Not completed — Death | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All baseline characteristics were analyzed on the safety analysis set which included all randomized participants who received at least one dose of DB study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Midazolam + SOC | Esketamine 28 mg + Placebo + SOC | Esketamine 56 mg + Placebo + SOC | Esketamine 84 mg + Placebo + SOC | Total
Number analyzed (Participants) | 63 | 29 | 31 | 23 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (1.45) | 14.9 (1.33) | 14.8 (1.52) | 14.3 (1.43) | 14.9 (1.46)
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 0 | 0 | 0 | 0 | 0
  Adolescents (12-17 years) | 63 | 29 | 31 | 23 | 146
  Adults (18-64 years) | 0 | 0 | 0 | 0 | 0
  From 65 to 84 years | 0 | 0 | 0 | 0 | 0
  85 years and over | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 24 | 25 | 17 | 114
  Male | 15 | 5 | 6 | 6 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 7 | 8 | 3 | 34
  Not Hispanic or Latino | 46 | 19 | 20 | 19 | 104
  Unknown or Not Reported | 1 | 3 | 3 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 2
  Asian | 1 | 0 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 4 | 1 | 4 | 15
  White | 53 | 25 | 23 | 17 | 118
  More than one race | 0 | 0 | 2 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Children's Depression Rating Scale-Revised (CDRS-R) Total Score at 24 Hours Post First Dose (Day 2)
Description: The CDRS-R is a validated 17- item, clinician-rated instrument developed to assess depressive symptomatology in children. Scores were based on interviews with both the child and their caregiver. Of the 17-item, 3 items were non-verbal behavior (listless speech, hypoactivity, and depressed affect) rated on a 5-point scale from 1 (no depression) to 5 (severe depression) and 14 items were rated on a 7-point scale from 1 (no depression) to 7 (severe depression), where higher score indicated more severe depression. The CDRS-R total score was the sum of the 17-tems score and it ranged from 17 (normal) to 113 (severe depression). Higher score indicated more severe depression and worse outcome.
Time Frame: Baseline (predose on Day 1) and 24 hours post first dose on Day 1 (i.e., Day 2)
Population: Full efficacy analysis set for DB phase included all randomized participants who received at least 1 dose of DB study medication during the DB phase and had both baseline & post dose evaluation for CDRS-R total score. As pre-planned in study statistical analysis plan (SAP), data were planned to be collected and analyzed on pooled population who had received esketamine (56 mg/84 mg) in arms "Esketamine 56 mg + Placebo + SOC" and "Esketamine 84 mg + Placebo + SOC" respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Pooled Esketamine 56 mg + Esketamine 84 mg: All participants who received intranasal doses of esketamine 56 mg nasal spray (2 doses in each nostril, 14 mg per spray + 1 dose of matched placebo nasal spray) and esketamine 84 mg nasal spray (3 doses in each nostril, 14 mg per spray) along with placebo matched to midazolam oral solution times per week for 4 weeks (i.e., on Days 1, 4, 8, 11, 15, 18, 22, and 25).
Arm/Group | Placebo + Midazolam + SOC | Esketamine 28 mg + Placebo + SOC | Esketamine 56 mg + Placebo + SOC | Esketamine 84 mg + Placebo + SOC | Pooled Esketamine 56 mg + Esketamine 84 mg
Number analyzed (Participants) | 63 | 28 | 31 | 23 | 54
Units on a scale | -26.2 (16.72) | -29.6 (18.15) | -31.8 (12.92) | -30.3 (17.48) | -31.2 (14.90)
Statistical Analysis 1: Comparison: Placebo + Midazolam + SOC vs Pooled Esketamine 56 mg + Esketamine 84 mg; A pooled (54 mg and 84 mg) sequential multiple testing procedure was implemented to control type I error by comparing pooled data against midazolam + placebo matched to esketamine nasal spray; Test type: Superiority; p = 0.037, ANCOVA — Threshold for significance for p-value was 0.05; Difference of LS Means = -5.8, 95% CI 2-sided [-11.19 to -0.35], Standard Error of Mean 2.74
Statistical Analysis 2: Comparison: Placebo + Midazolam + SOC vs Esketamine 84 mg + Placebo + SOC; Individual esketamine dose (84 mg versus medazolam + esketamine matched placebo) independent testing was planned to be performed after pooled (56 mg + 84 mg) analysis; Test type: Superiority; p = 0.123, ANCOVA — Threshold for significance for p-value was 0.05; Difference of LS Mean = -5.7, 95% CI 2-sided [-12.91 to 1.55], Standard Error of Mean 3.65
Statistical Analysis 3: Comparison: Placebo + Midazolam + SOC vs Esketamine 56 mg + Placebo + SOC; Individual esketamine dose (56 mg versus medazolam + esketamine matched placebo) independent testing was planned to be performed after pooled (56 mg + 84 mg) analysis; Test type: Superiority; p = 0.072, ANCOVA — Threshold for significance for p-value was 0.05; Difference of LS Means = -5.9, 95% CI 2-sided [-12.25 to 0.53], Standard Error of Mean 3.23
Statistical Analysis 4: Comparison: Placebo + Midazolam + SOC vs Esketamine 28 mg + Placebo + SOC; Test type: Superiority; Difference of LS Means = -2.4, 95% CI 2-sided [-9.08 to 4.19], Standard Error of Mean 3.35

ADVERSE EVENTS:
Time Frame: Double Blind treatment phase: From Day 1 to Day 25; Follow-up phase: From Day 26 up to end of post-treatment follow-up phase (Day 200)
Description: Safety analysis set for DB treatment phase included all randomized participants who received at least 1 dose of study medication during the DB treatment phase. Follow-up analysis set for follow-up phase included all participants who completed the DB treatment phase and either entered the follow-up phase or had provided AE data after the DB treatment phase.
Groups:
- DB: Placebo + Midazolam + SOC: In the double blind (DB) phase, participants received 3 intranasal doses of placebo (matched to esketamine nasal spray) using 3 devces, each device at time points 0, 5 and 10 minutes (min) respectively. For each device, 1 spray was administered into each nostril (that is total of 2 sprays/device). An oral solution of midazolam 0.125 milligrams per kilogram (mg/kg) was administered immediately before the first intranasal dose. Study drugs were taken 2 times per week for 4 weeks (on Days 1, 4, 8, 11, 15, 18, 22, and 25). During the study, all participants were treated with Standard of care (SOC): antidepressant treatment (either fluoxetine or escitalopram or sertaline) based on clinical judgement, initiated, or optimized on Day 1 or up to 7 days after first dose of study drug administration (on Day 1), if starting two medications simultaneously was not consistent with local clinical practice, and psychotherapy. After DB treatment phase, participants entered post-treatment FU phase and received no study drug.
- DB: Esketamine 28 mg + Placebo + SOC: In DB phase, participants received 1 intranasal dose of esketamine 28 mg nasal spray using a device, at 0 min, followed by 2 intranasal doses of placebo (matched to esketamine) using 2 devices, 1 at 5 min and another at 10 min, respectively. For each device, 1 spray (esketamine 14 mg/placebo) was administered into each nostril (that is total of 2 sprays = esketamine 28 mg/placebo). Placebo oral solution (matched to midazolam 0.125 mg/kg) was administered immediately before first intranasal dose. Study drugs were taken 2 times per week for 4 weeks (on Days 1, 4, 8, 11, 15, 18, 22, and 25). During study, all participants received SOC: antidepressant treatment (fluoxetine or escitalopram or sertaline) based on clinical judgement, initiated or optimized on Day 1 or up to 7 days after first dose (on Day 1), if starting two medications simultaneously was not consistent with local clinical practice, and psychotherapy. After DB phase, participants entered post-treatment FU phase and received no study drug.
- DB: Esketamine 56 mg + Placebo + SOC: In DB phase, participants received 2 intranasal doses of esketamine 56 mg nasal spray using 2 devices, 1 at 0 min and another at 5 min, followed by 1 intranasal dose of placebo (matched to esketamine) using 1 device at 10 min. For each device, 1 spray (esketamine 14 mg/placebo) was administered into each nostril (that is total of 2 sprays = esketamine 28 mg/placebo). Placebo oral solution (matched to midazolam 0.125 mg/kg) was administered immediately before first intranasal dose. Study drugs were taken 2 times per week for 4 weeks (on Days 1, 4, 8, 11, 15, 18, 22, and 25). During study, all participants received SOC:antidepressant treatment (fluoxetine or escitalopram or sertaline) based on clinical judgement, initiated or optimized on Day 1 or up to 7 days after first dose (on Day 1), if starting two medications simultaneously was not consistent with local clinical practice, and psychotherapy. After DB phase, participants entered post-treatment FU phase and received no study drug.
- DB: Esketamine 84 mg + Placebo + SOC: In DB phase, participants received 3 intranasal doses of esketamine 84 mg nasal spray using 3 devices, each device at time points 0, 5 and 10 minutes respectively. For each device, 1 spray (esketamine 14 mg/placebo) was administered into each nostril (that is total of 2 sprays = esketamine 28 mg/placebo). Placebo oral solution (matched to midazolam 0.125 mg/kg) was administered immediately before first intranasal dose. Study drugs were taken 2 times per week for 4 weeks (on Days 1, 4, 8, 11, 15, 18, 22, and 25). During study, all participants received SOC:antidepressant treatment (fluoxetine or escitalopram or sertaline) based on clinical judgement, initiated or optimized on Day 1 or up to 7 days after first dose (on Day 1), if starting two medications simultaneously was not consistent with local clinical practice, and psychotherapy. After DB phase, participants entered post-treatment FU phase and received no study drug.
- FU Phase: Placebo + Midazolam + SOC; FU Phase: Esketamine 28 mg + Placebo + SOC; FU Phase: Esketamine 84 mg + Placebo + SOC: After completion of DB treatment phase, participants entered post-treatment follow-up phase and received no study drug. During the study, all participants were treated with SOC: antidepressant treatment (either fluoxetine or escitalopram or sertaline) based on clinical judgement, initiated or optimized on Day 1 or up to 7 days after 1st dose of study drug administration (on Day 1), if starting two medications simultaneously was not consistent with local clinical practice, and psychotherapy.
- FU Phase: Esketamine 56 mg + Placebo + SOC: After completion of DB treatment phase, participants entered post-treatment follow-up phase and received no study drug. During the study, all participants were treated with SOC: antidepressant treatment (either fluoxetine or escitalopram or sertaline) based on clinical judgement, initiated or optimized on Day 1 or up to 7 days after 1st dose of study drug administration (on Day 1), if starting two medications simultaneously was not consistent with local clinical practice, and psychotherapy.).
Arm/Group | DB: Placebo + Midazolam + SOC | DB: Esketamine 28 mg + Placebo + SOC | DB: Esketamine 56 mg + Placebo + SOC | DB: Esketamine 84 mg + Placebo + SOC | FU Phase: Placebo + Midazolam + SOC | FU Phase: Esketamine 28 mg + Placebo + SOC | FU Phase: Esketamine 56 mg + Placebo + SOC | FU Phase: Esketamine 84 mg + Placebo + SOC
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/29 | 0/31 | 0/23 | 1/59 | 0/29 | 0/29 | 0/21
Serious Adverse Events (participants affected / at risk) | 9/63 | 4/29 | 7/31 | 1/23 | 19/59 | 10/29 | 8/29 | 7/21
Other Adverse Events (participants affected / at risk) | 57/63 | 26/29 | 30/31 | 23/23 | 48/59 | 21/29 | 19/29 | 14/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB: Placebo + Midazolam + SOC (N=63) | DB: Esketamine 28 mg + Placebo + SOC (N=29) | DB: Esketamine 56 mg + Placebo + SOC (N=31) | DB: Esketamine 84 mg + Placebo + SOC (N=23) | FU Phase: Placebo + Midazolam + SOC (N=59) | FU Phase: Esketamine 28 mg + Placebo + SOC (N=29) | FU Phase: Esketamine 56 mg + Placebo + SOC (N=29) | FU Phase: Esketamine 84 mg + Placebo + SOC (N=21)
HIV Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Humerus Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food Refusal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychomotor Hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Status Migrainosus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bipolar Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Completed Suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depression Suicidal (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (2)
Intentional Self-Injury (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Major Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 3 (3) | 3 (3) | 2 (2) | 0 (0) | 4 (4) | 5 (10) | 3 (3) | 3 (6)
Suicide Attempt (Psychiatric disorders) | 5 (6) | 1 (1) | 5 (5) | 1 (1) | 9 (11) | 3 (3) | 5 (11) | 4 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB: Placebo + Midazolam + SOC (N=63) | DB: Esketamine 28 mg + Placebo + SOC (N=29) | DB: Esketamine 56 mg + Placebo + SOC (N=31) | DB: Esketamine 84 mg + Placebo + SOC (N=23) | FU Phase: Placebo + Midazolam + SOC (N=59) | FU Phase: Esketamine 28 mg + Placebo + SOC (N=29) | FU Phase: Esketamine 56 mg + Placebo + SOC (N=29) | FU Phase: Esketamine 84 mg + Placebo + SOC (N=21)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 2 (2) | 2 (5) | 2 (7) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 1 (8) | 2 (3) | 4 (7) | 3 (12) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 4 (5) | 3 (3) | 2 (2) | 3 (5) | 7 (8) | 1 (1) | 2 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (3) | 6 (7) | 1 (1) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 (0) | 6 (19) | 6 (29) | 5 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (13) | 8 (19) | 15 (43) | 13 (37) | 9 (10) | 3 (3) | 3 (11) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5) | 5 (5) | 7 (11) | 6 (7) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (9) | 1 (4) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Feeling Drunk (General disorders) | 2 (2) | 1 (6) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Weight Increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 4 (4) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 27 (44) | 16 (76) | 16 (88) | 16 (58) | 3 (5) | 0 (0) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 15 (53) | 10 (57) | 8 (33) | 9 (39) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 18 (33) | 10 (17) | 13 (34) | 7 (18) | 12 (20) | 10 (14) | 7 (11) | 3 (6)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 5 (12) | 8 (24) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory Impairment (Nervous system disorders) | 4 (6) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (2) | 2 (3) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 9 (45) | 2 (2) | 4 (7) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 24 (123) | 10 (36) | 9 (34) | 8 (25) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 1 (3)
Tremor (Nervous system disorders) | 1 (1) | 3 (4) | 2 (2) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 2 (3) | 1 (4) | 1 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 10 (15) | 3 (3) | 4 (5) | 2 (6) | 7 (16) | 3 (6) | 4 (4) | 3 (11)
Confusional State (Psychiatric disorders) | 4 (12) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 4 (5)
Disinhibition (Psychiatric disorders) | 0 (0) | 2 (8) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dissociation (Psychiatric disorders) | 11 (24) | 12 (46) | 12 (51) | 11 (58) | 1 (1) | 1 (1) | 1 (4) | 0 (0)
Euphoric Mood (Psychiatric disorders) | 6 (12) | 6 (17) | 5 (22) | 5 (24) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination, Visual (Psychiatric disorders) | 3 (7) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Illusion (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Initial Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 8 (16) | 4 (4) | 2 (7) | 2 (3) | 1 (1) | 4 (4) | 2 (3) | 0 (0)
Intentional Self-Injury (Psychiatric disorders) | 12 (19) | 6 (9) | 6 (12) | 5 (7) | 21 (33) | 7 (19) | 3 (3) | 7 (17)
Suicidal Ideation (Psychiatric disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 2 (3) | 0 (0) | 2 (2)
Time Perception Altered (Psychiatric disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 3 (6) | 0 (0) | 1 (1) | 1 (1) | 4 (9) | 0 (0) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (5) | 3 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 2 (2) | 3 (5) | 3 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (4) | 1 (1) | 2 (2) | 2 (2) | 2 (3) | 0 (0) | 1 (1)
Pharyngeal Hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (4) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (9) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-11-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT03185819/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT03185819/SAP_001.pdf